CLINICAL TRIAL: NCT04209231
Title: Principal Investigator
Brief Title: Effect of Vitamin D on Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hatice Yemenoğlu, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: RecepTayyipErdoganUniversity
Record Dates: First submitted 2019-12-07; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Vitamin D Deficiency; Periodontal Diseases
Keywords: periodontitis; gingivitis; vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Periodontal Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chronic periodontitis
  Interventions: Other: 1.25(OH)2D3; Other: 25(OH)D
- chronic gingivitis
  Interventions: Other: 1.25(OH)2D3; Other: 25(OH)D
- periodontally healthy
  Interventions: Other: 1.25(OH)2D3; Other: 25(OH)D

INTERVENTIONS:
Other: 1.25(OH)2D3
Other: 25(OH)D

SUMMARY:
Background. Vitamin D has both direct effects on bone metabolism and an antimicrobial effect on periodontopathogens. It also inhibits inflammatory mediators that contribute to periodontal destruction. The purpose of this study was to evaluate the association between serum 1.25-hydroxyvitamin D (1.25(OH)2D3) and 25(OH)D levels and periodontal inflammation.

Methods. This study included 28 subjects with chronic gingivitis, 29 subjects with chronic periodontitis and 25 periodontally healthy subjects. Blood samples were collected from the participants to determine serum levels of 25(OH)D, 1.25(OH)2D3, tumour necrosis factor α (TNF-α), C-reactive protein (CRP) and interleukin 6 (IL-6). Clinical parameters were recorded. Results were statistically analysed with a Shapiro-Wilk's test, Mann-Whitney U test, Kruskal-Wallis H test, Wilcoxon test and post-hoc multiple comparison test.

DETAILED DESCRIPTION:
The subjects included in the study were selected from among patients who applied to our clinic, for routine periodontal examinations. Individuals who had been using immunosuppressive drugs and antibiotics for the past three months, smokers, individuals who had periodontal treatment within the past six months, and individuals with additional or supplementary vitamin D and systemic diseases were excluded from the study. In addition, since the region's level of sunlight exposure may have an effect on the level of vitamin D, participants were required to live in the region for the last five years.

A total of 82 subjects, including 25 as a periodontally healthy control group, 28 with chronic gingivitis and 29 with chronic periodontitis, were included in the study. Clinical criteria for chronic periodontitis are the formation of plaque and calculus and ≥ 5 milimeter (mm) pocket depth or attachment loss in more than 30% of the teeth. Diagnosis criteria for chronic gingivitis are the formation of plaque and/or calculus in the mouth, bleeding, and no loss of pocket or attachment. The diagnosis criteria for periodontally healthy individuals are having clinically healthy periodontal tissues or minimal periodontal inflammation, with no loss of pocket or attachment.

ELIGIBILITY:
Inclusion Criteria:

* live in the region for the last five years.

Exclusion Criteria:

* individuals who had been using immunosuppressive drugs and antibiotics for the past three months, smokers, individuals who had periodontal treatment within the past six months, and individuals with additional or supplementary vitamin D and systemic diseases.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: live in the region for the last five years.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
periodontal paremeters | December 2015- March 2016
  Attachment loss and pocket depth were measured from the six surfaces of the teeth (buccal, palatal/lingual, mesiobuccal, mesiolingual, distobuccal and distolingual) except for the third molars. These values were calculated in millimeters (mm).
laboratory analysis | December 2015- March 2016
  Venous blood samples were collected from the patients on the examination day that were allowed to rest for half an hour and then centrifuged at 4000 rpm for 10 min. Serum samples were separated into Eppendorf tubes and stored at -20°C until the experiment day. On the day of biochemical analysis, serum samples were thawed at room temperature and studied according to the manufacturer's instructions. TNF-a, 1,25(OH)2D3, IL-6 were calculated in pg/mL, 25(OH)D was calculated ng/mL and CRP was calculated mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No